CLINICAL TRIAL: NCT00928837
Title: A Double-Blind,Randomized, Placebo Controlled, Parallel Group, Multi-Center Study of Flavocoxid (Limbrel) Versuss Naproxen in Subjects With Moderate-Severe Osteoarthritis of the Knee
Brief Title: Study of Flavocoxid (Limbrel) Versus Naproxen in Subjects With Moderate-Severe Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Primus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Primus Pharmaceuticals LOA-03P
Record Dates: First submitted 2008-11-12; First posted 2009-06-26 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2009-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — flavocoxid; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- flavocoxid 250 mg (Active Comparator): Medical Food product
  Interventions: Other: flavocoxid 250 mg
- Naproxen (Active Comparator): antiinflammatory
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- flavocoxid 500 mg (Experimental): medical food product
  Interventions: Dietary Supplement: Flavocoxid 500 mg

INTERVENTIONS:
Dietary Supplement: Flavocoxid 500 mg — flavonoid mixture
  Other Names: Limbrel 500 mg
  Arms: flavocoxid 500 mg
Drug: Naproxen — non-steroidal anti-inflammatory drug
  Other Names: naprosyn
  Arms: Naproxen
Other: Placebo — Placebo
  Arms: Placebo
Other: flavocoxid 250 mg — Medical food product
  Other Names: Limbrel 250 mg
  Arms: flavocoxid 250 mg

SUMMARY:
The purpose of the study is to compare the efficacy and safety of flavocoxid (Limbrel) with Naproxen and placebo in OA of the knee.

DETAILED DESCRIPTION:
To compare the efficacy, safety, quality of life and economic impact of flavocoxid vs naproxen.

ELIGIBILITY:
Inclusion Criteria:Major inclusión criteria:

1. Adults of either gender, ages 35-85, in general good health
2. Diagnosed with OA of the knee, K-L Grade 2-3
3. History of positive response to NSAID's or COX-2 inhibitors
4. Able and willing to discontinue other medicinal OA therapies for length of the study (subjects may continue low dose aspirin for cardioprotection)
5. Females of child bearing potential must use acceptable method of birth control

Major exclusion criteria:

1. Unwilling or unable to read and sign informed consent document
2. Pregnant and nursing women
3. History of severe cardiovascular disease including, but not limited to chronic angina, congestive heart failure, uncontrolled hypertension, acute myocardial infarction within past year
4. K-L grade 1 or 4 OA of the target knee
5. chronic bleeding disorder or present use of anticoagulants
6. History of upper G-I bleed in the past 5 years
7. Significant renal disease including nephrotic syndrome, proteinuria >1 gm/24 hrs or serum Creatinine >2.0
8. Any arthritic disease that is or has the potential to affect the knees during the course of the study
9. Any other condition that might confound evaluation of the target joint including, but not limited to, bursitis, tendonitis or internal derangement in or about the knee, gait disturbances (e.g. mechanical, neurological conditions or disorders of the back), fibromyalgia, polyneuropathies, etc.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-03; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
to compare the efficacy of 2 doses of flavocoxid with that of naproxen and placebo at 12 weeks | 3 months
  comparison of short WOMAC and timed walk
to compare the safety of 2 doses of flavocoxid with that of naproxen and placebo at 12 weeks | 3 months
  Comparison of FS-36, subject tolerability VAS

SECONDARY OUTCOMES:
to compare the efficacy of 2 doses of flavocoxid with that of naproxen and placebo at 12 weeks | 6 months
  comparison of short WOMAC and timed walk
to compare the safety of 2 doses of flavocoxid with that of naproxen and placebo at 12 weeks | 6 months
  Comparison of FS-36, subject tolerability VAS

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Kivitz, MD, Principal Investigator — Recruiting Altoona Center for Clinical Research 1125 Old Rt 220 North Duncansville PA 16635 Phone 814-693-0300 Fax 814-693-0400; Timothy S Truitt, MD, Principal Investigator — Recruiting MIMA Century Research Associates 65 E. Nasa Blvd Suite 106 Melbourne FL 32901 Phone 321-723-1203 Fax 321-725-3602; Joy Schechtman, DO, Principal Investigator — Sun Valley Arthritis Ltd. 6525 W. Sack Drive Suite 108 Glendale AZ 85308 Phone 623-825-5591 Fax 623-362-9264; David S Silver, MD, Principal Investigator — 8691 Wilshire Blvd Suite 301 Beverly Hills CA 90211 phone 310-657-9650 Fax 310-659-2841; Nathan Wei, MD, Principal Investigator — Arthritis and Osteoporosis Center of Maryland71 Thomas Johnson Drive Frederick MD 21702 Phone 301-694-5800 Fax 301 694-0187; Norman B Gayliss, MD, Principal Investigator — 2845 Aventura Blvd. Suite 100 Aventura FL 33180 Phone 305-932-4295 Fax 305-932-6335; David A. McLain, MD, Principal Investigator — 2022 Brookwood Medical Center Drive Suite 211 Birmingham AL 35209 Phone 205-877-2555 Fax 205-877-2790
Locations (1):
- Alan Kivitz MD, Duncansville, Pennsylvania, United States

REFERENCES:
- See also: Primus Pharmaceuticals,Inc. — http://www.primusrx.com